CLINICAL TRIAL: NCT05671263
Title: Genital Lichen Sclerosus - Epidemiology, Comorbidities and the Role of Vulvar and Penile Microbiome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Jönköping County (Other Government)
Collaborators: FORSS, Forskningsrådet i Sydöstra Sverige (Unknown); Futurum - Academy for health and care (Unknown)
Responsible Party: Principal Investigator, Sandra Jerkovic Gulin, Principal Investigator, Region Jönköping County
Other Study IDs: EPM 2020-xxxxx
Record Dates: First submitted 2022-01-14; First posted 2023-01-04 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Lichen Sclerosus
Keywords: lichen sclerosus; penis cancer; vulva cancer
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus; Penile Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cotton swab sample will be taken from a penile lesional skin in men with genital LSc before treatment and from vulvar lesional skin in women with genital LSc before treatment and after the treatment. The same procedure with healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- cases women LSc: women with LSc- vulvar lesional skin (including mons pubis, labia minora and labia majora) in women with genital LSc
- cases men LSc: men with LSc -penile lesional skin (including glans penis and coronal sulcus) in men with genital LSc
- control women: women without genital disease
- control men: men without genital disease

SUMMARY:
In genital LSc, three pathological processes are implicated in disease development: inflammation, sclerosis/fibrosis and neoplasia. The role of genital microbiome is still to be investigated and explained. Genital LSc microbiome studies are missing. The ecological community of microorganisms that are present on our body and of the body itself defines the human skin microbiome. Revealing the genital microbiome may potentially lead to new therapies of genital LSc. The primary aim is to analyze genital microbiome before and after the treatment (topical corticosteroids or topical calcineurin inhibitors or circumcision) in both male and female patients diagnosed with genital LSc as well as to analyze genital microbiome in healthy (non-genital LSc) controls. 2) The secondary aim is to determine incidence and prevalence of male and female genital LSc in Sweden and its association with other diseases. The Study will be divided in two parts

1. PART A: Prospective case control study on the effect of treatment on the genital skin microbiome of patients with genital LSc and on the role of genital microbiome in treatment resistance of genital LSc
2. PART B: Swedish nationwide register-based cohort study to analyse incidence, prevalence and comorbidities of genital LSc

DETAILED DESCRIPTION:
PART A: Microbiome study The participants will be included continuously at the Dermatology clinic in connection with the regular doctor's visit. All cases included will be asked to complete Dermatology Life Quality Index (DLQI) questionnaires. A first cotton swab sample will be taken from a penile affected skin (including glans penis and coronal sulcus) in men with genital LSc before treatment and from vulvar affected skin (including mons pubis, labia minora and labia majora) in women with genital LSc before treatment. A second cotton swab sample will be taken from the same sites at week 12 after the treatment including both topical therapies and circumcision. The topical treatment will be discontinued a week prior to visit. Allowed treatment options include topical and systemic corticosteroids and topical calcineurin inhibitors (tacrolimus, pimecrolimus) for both sexes and circumcision for men. In extreme resistant cases of genital LSc in women even methotrexate, hydroxychloroquine will be recommended as systemic treatment. The samples will be analyzed using 16S ribosomal RNA metagenomic sequencing to identify the microbiome. Microbio analysis at Laboratory Medicine, Ryhov is today an established method based on "next generation sequencing" (NGS) for analysis of 16S rDNA, which has previously been used for analysis of skin and throat samples in psoriasis projects as well as intestinal biopsies and faecal samples from patients with inflammatory bowel disease. The microbial skin flora is sampled using a microbial swab (eNAT, Copan). Taxonomic classification and a determination of numbers per sample of each taxonomic unit is made on the basis of a reference database (Silva; https://www.arb-silva.de/) and suitable bioinformatics analysis tools such as QIIME2 (https://qiime2.org/) and mothur (https://mothur.org/). Group differences are examined with generalized linear models adapted for number data (eg DESeq2 and glue; https://bioconductor.org/) in the statistical programming environment R (https://cran.r-project.org/), and the analyzes are corrected based on gender and age. The biochemical properties of the microbiome are predicted using reference genomes based on the 16S composition of the samples using PICRUSt2 (https://github.com/picrust/picrust2/wiki), and examined for group differences.

PART B:

* A retrospective nationwide cohort study will be conducted using national Swedish registers (National Patient Register, Swedish Cancer Register) and LISA database (Longitudinal integration database for health insurance and labor market studies). The patients diagnosed with LSc (ICD-10 diagnosis code - L90) during 20-years period between January 1, 2001 and January 1, 2021 will be selected.
* Comorbidity will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Genital LSc diagnosed by a dermatologist (cases) and individuals without genital LSc (controls)

Exclusion Criteria:

* Age under 18
* Pregnancy
* Current diagnosis of cancer or ongoing treatment for cancer (not applicable for basal cell carcinoma (BCC) and squamous cell carcinoma (SCC) of extra-genital localization)
* Male patients already underwent circumcision as LSc treatment before inclusion into the study
* Ongoing systemic anti-inflammatory and/or immunomodulating treatment or having discontinued such treatment within the last week
* Ongoing treatment with systemic antibiotics or having discontinued such treatment within the last week
* Treatment with topical antibiotics, topical corticosteroids and/or topical calcineurin inhibitors (tacrolimus, pimecrolimus) on the sampling area within the last week
* Having used antiseptics and disinfectants on the sampling area 24 hours prior to the samples being taken
* Persons not understanding Swedish or not being able to leave consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Genital LSc diagnosed by a dermatologist (cases) and individuals without genital LSc (controls). Adults only.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life in patients with genital lichen sclerosus (The Dermatology Life Quality Index -DLQI) | 24 months
  DLQI questionnaire data will be analysed, the DLQI score will be calculated 0-30 (higher the score, more effect on patient´s quality of life)
The role of genital microbiome in the treatment resistance of genital LSc | 24 months
  analysis of genital microbiome will be performed, 16S ribosomal RNA metagenomic sequencing will be conducted on samples.
Lichen slerosus comorbidity will be determined in a register study | 24 months
  A retrospective nationwide cohort study will be conducted using national Swedish registers (National Patient Register, Swedish Cancer Register) and LISA database (Longitudinal integration database for health insurance and labor market studies). The patients diagnosed with LSc (ICD-10 diagnosis code - L90) during 20-years period between January 1, 2001 and January 1, 2021 will be selected

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Seifert, PhD AssProf, Study Chair — Länssjukhuset Ryhov, Hudkliniken; Jan Söderman, PhD AssProf, Study Chair — Länssjukhuset Ryhov, Division of Microbiology; sandra j gulin, PhD, Principal Investigator — Länssjukhuset Ryhov, Hudkliniken; Annika Bergman, PhD, Study Chair — Länssjukhuset Ryhov, Division of Microbiology; Linda Berglind, Study Chair — Länssjukhuset Ryhov, Division of Microbiology; Charlotta Enerbäck, PhD Prof, Study Chair — Department of Biomedical and Clinical Sciences, Faculty of Health Sciences, Linköping University
Locations (1):
- Department of Dermatology Ryhov County Hospital (Hudkliniken Länssjukhus Ryhov), Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: No
results will be published